CLINICAL TRIAL: NCT01190436
Title: A Study on the Efficacy of Bisoprolol and Its Influence on Selected Biochemical Parameters in Filipino Hypertensive Patients With Diabetes
Brief Title: A 12-week, Multicentric Study to Evaluate the Safety and Efficacy of Bisoprolol in Filipino Hypertensive Subjects With Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Inc., Philippines (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200006-512
Record Dates: First submitted 2010-08-26; First posted 2010-08-27 (Estimated); Results first posted 2014-05-23 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Hypertension
Keywords: Hypertension; Diabetes Mellitus; Bisoprolol
MeSH Terms: conditions — Hypertension; Diabetes Mellitus | interventions — Bisoprolol; bisoprolol, hydrochlorothiazide drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bisoprolol (Experimental)
  Interventions: Drug: Bisoprolol

INTERVENTIONS:
Drug: Bisoprolol — Bisoprolol will be administered at an initial dose of 5 milligram (mg) once daily for 2 weeks. If the blood pressure would be greater than or equal to 130/80 mmHg after 2 weeks, then dose will be adjusted to 10 mg once daily. Total duration of study treatment will be 12 weeks.
  Other Names: Bisoprolol fumarate, Ziac

SUMMARY:
The aim of this 12-week, multicenter, interventional, prospective, open-label and single-arm study is to evaluate the safety and efficacy of 5 milligram per day (mg/day) and 10 mg/day bisoprolol in Filipino hypertensive subjects with diabetes as monotherapy or as an add-on therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects with hypertension, either newly diagnosed or treated but currently uncontrolled as defined by Joint National Committee (JNC) 7 for subjects with Type 2 diabetes mellitus (T2DM) (that is, greater than or equal to [>=] 130/80 mmHg)
* Aged at least 18 years old
* Diagnosed with T2DM and already on anti-diabetic therapy, and with glycosylated hemoglobin of less than 7 percent

Exclusion Criteria:

* Subjects who were already on beta-blocker therapy at the time of recruitment
* Subjects with heart rate of at most 60 beats per minute (bpm) at rest
* Subjects with secondary hypertension, congenital heart disease, coronary artery disease, peripheral arterial disease or congestive heart failure in any stage
* Subjects with coronary conduction disorders (bundle branch block)
* Subjects with signs of definitive target organ damage consistent with World Health Organization (WHO) Stage III or with severe renal or hepatic disease
* Subjects who are pregnant or expect to be pregnant within the 24-week study period
* Subjects on oral contraceptives
* Subjects with asthma or a history of asthma
* Subjects with documented severe renal disease
* Subjects on anti-neoplastic drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2009-12; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Inc., Philippines
Locations (1):
- Research Site, Manila, Philippines

RESULTS

PARTICIPANT FLOW:
Groups:
- Bisoprolol: Bisoprolol was administered at an initial dose of 5 milligram (mg) once daily for 2 weeks. If the blood pressure was greater than or equal to 130/80 millimeter of mercury (mmHg) after 2 weeks, then the dose was adjusted to 10 mg once daily. Total duration of study treatment was 12 weeks.
Period: Overall Study
Arm/Group | Bisoprolol
Started | 125
Completed | 86
Not Completed | 39
Not completed — Lost to Follow-up | 35
Not completed — Other | 4

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all participants who received at least 1 dose of study drug.
Arm/Group | Bisoprolol
Number analyzed (Participants) | 125
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.5 (12.1)
Gender [Count of Participants; unit: Participants]
  Female | 73
  Male | 52

OUTCOME MEASURES:

1. Secondary Outcome: Percentage of Participants With Increased Glycosylated Hemoglobin (HbA1c) at Week 12
Description: HbA1c represents the percentage of glycosylated hemoglobin. Percentage of participants with increased HbA1c (greater than 0.5% from baseline) at Week 12 was reported.
Time Frame: Week 12
Population: ITT population included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Bisoprolol
Number analyzed (Participants) | 125
percentage of participants | 16.8 (0.6)

2. Secondary Outcome: Mean Change From Baseline in HbA1c at Week 12
Description: HbA1c represents the percentage of glycosylated hemoglobin. The change in HbA1c at Week 12 was calculated as HbA1c at Week 12 minus HbA1c at baseline.
Time Frame: Baseline, Week 12
Population: ITT population included all participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: Percent HbA1c
Arm/Group | Bisoprolol
Number analyzed (Participants) | 125
Percent HbA1c
  Baseline | 6.28 (0.43)
  Change at Week 12 | 0.02 (0.59)

3. Primary Outcome: Mean Change From Baseline in Systolic and Diastolic Blood Pressure (BP) at Week 12
Description: The change in diastolic and systolic BP at Week 12 was calculated as diastolic and systolic BP at Week 12 minus diastolic and systolic BP at baseline, respectively.
Time Frame: Baseline, Week 12
Population: Intent-to-treat (ITT) population included all participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Bisoprolol
Number analyzed (Participants) | 125
mmHg
  Systolic BP: Baseline | 151.7 (20.1)
  Systolic BP: Change at Week 12 | 12.54 (18.39) [10.29 to 16.80]
  Diastolic BP: Baseline | 87.6 (8.2)
  Diastolic BP: Change at Week 12 | 8.48 (10.01) [6.71 to 10.25]

4. Primary Outcome: Percentage of Participants With Controlled BP
Description: Controlled BP was defined as BP less than 130/80 mmHg.
Time Frame: Week 12
Population: ITT population included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Bisoprolol
Number analyzed (Participants) | 125
percentage of participants | 42.4

5. Primary Outcome: Percentage of Participants With Response to Study Drug
Description: Response to study drug was defined as lowering of systolic BP by at least 10 mmHg from baseline.
Time Frame: Week 12
Population: ITT population included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Bisoprolol
Number analyzed (Participants) | 125
percentage of participants | 44.0

6. Primary Outcome: Mean Change From Baseline in Heart Rate at Week 12
Description: The change in heart rate at Week 12 was calculated as the heart rate at Week 12 minus heart rate at baseline.
Time Frame: Baseline, Week 12
Population: ITT population included all participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Bisoprolol
Number analyzed (Participants) | 125
beats per minute (bpm)
  Baseline | 78.2 (9.2)
  Change at Week 12 | 8.55 (9.24)

7. Secondary Outcome: Percentage of Participants With Increased Fasting Blood Sugar (FBS) at Week 12
Description: Percentage of participants with increased FBS (greater than 16 milligram per deciliter [mg/dL] from baseline) at Week 12 was reported.
Time Frame: Week 12
Population: ITT population included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Bisoprolol
Number analyzed (Participants) | 125
percentage of participants | 15.2

8. Secondary Outcome: Mean Change From Baseline in Fasting Blood Sugar (FBS) Level at Week 12
Description: The change in FBS level at Week 12 was calculated as FBS level at Week 12 minus FBS level at baseline.
Time Frame: Baseline, Week 12
Population: ITT population included all participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Bisoprolol
Number analyzed (Participants) | 125
mg/dL
  Baseline | 117.1 (25.8)
  Change at Week 12 | -5.49 (25.83)

9. Primary Outcome: Percentage of Participants With Decrease in Heart Rate by at Least 10 Bpm at Week 12
Time Frame: Week 12
Population: ITT population included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Bisoprolol
Number analyzed (Participants) | 125
percentage of participants | 36.8

10. Secondary Outcome: Mean Change From Baseline in Total Cholesterol, Low Density Lipoprotein (LDL) Cholesterol, High Density Lipoprotein (HDL) Cholesterol and Triglyceride Level at Week 12
Description: The change in total cholesterol, LDL cholesterol, HDL cholesterol and triglyceride level at Week 12 was calculated as total cholesterol, LDL cholesterol, HDL cholesterol and triglyceride level at Week 12 minus total cholesterol, LDL cholesterol, HDL cholesterol and triglyceride level at baseline, respectively.
Time Frame: Baseline, Week 12
Population: ITT population included all participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Bisoprolol
Number analyzed (Participants) | 125
mg/dL
  Total cholesterol: Baseline | 183.7 (39.7)
  Total cholesterol: Change at Week 12 | 1.25 (32.14)
  LDL cholesterol: Baseline | 105.5 (31.0)
  LDL cholesterol: Change at Week 12 | -1.20 (22.40)
  HDL cholesterol: Baseline | 52.0 (15.6)
  HDL cholesterol: Change at Week 12 | 0.88 (12.23)
  Triglyceride: Baseline | 122.8 (55.2)
  Triglyceride: Change at Week 12 | 2.59 (38.32)

11. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An adverse event (AE) was defined as any new untoward medical occurrences/worsening of pre-existing medical condition without regard to possibility of causal relationship.
Time Frame: Baseline up to Week 12
Population: ITT population included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Groups:
- Bisoprolol: Bisoprolol was administered at an initial dose of 5 milligram (mg) once daily for 2 weeks. If the blood pressure was greater than 130/80 millimeter of mercury (mmHg) or equal to 130/80 mmHg after week, bisoprolol dose adjusted to 10 mg once daily. Duration of the treatment was 12 weeks.
Arm/Group | Bisoprolol
Number analyzed (Participants) | 125
participants | 8

ADVERSE EVENTS:
Time Frame: Baseline up to Week 12
Description: Serious Adverse event (SAE): Any AE that resulted in death; was life threatening; resulted in persistent/significant disability/incapacity; resulted in/prolonged an existing in-patient hospitalization; was a congenital anomaly/birth defect; or was a medically important condition.
Arm/Group | Bisoprolol
Serious Adverse Events (participants affected / at risk) | 0/125
Other Adverse Events (participants affected / at risk) | 8/125
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bisoprolol (N=125)
Hypersensitivity (Immune system disorders) | 1
Chest pain (General disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 1
Headache (Nervous system disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Palpitations (Cardiac disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Dizziness (Nervous system disorders) | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI shall make no press release, advertising or other promotional written or oral statements to public in connection with any reference to Sponsor's name of any member of Sponsor's staff, or PI, without prior approval of Sponsor or designated agent.

PI and/or Co-I shall not publish any information related to study data/results without first obtaining prior written consent of Sponsor and agrees to submit to Sponsor for review, a copy of any proposed publication resulting from completed study.